CLINICAL TRIAL: NCT04301115
Title: Attachment-retained Unilateral Partial Denture Versus Tooth Implant Supported Prosthesis in Mandibular Distal Extension Cases
Brief Title: Unilateral Attachment Versus Tooth Implant Supported Bridge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sharaf Mohamed Yahia, lecturer of prosthodontics, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 201802
Record Dates: First submitted 2020-03-02; First posted 2020-03-10 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Edentulous Jaw
Keywords: attachment,; patient satisfaction; radiographic evaluation; implant
MeSH Terms: conditions — Jaw, Edentulous; Patient Satisfaction | interventions — Congresses as Topic; Denture, Partial

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- conventional group (Active Comparator): conventional partial denture
  Interventions: Other: CONVENTIONAL
- attachment group (Experimental): unlateral attachment retained partial denture
  Interventions: Other: attachment
- tooth implant supporeted prosthesis (Experimental): tooth implant supported bridge
  Interventions: Other: bridge

INTERVENTIONS:
Other: attachment — unilateral attachment from rehine 83
  Arms: attachment group
Other: bridge — tooth implant supported bridge
  Arms: tooth implant supporeted prosthesis
Other: CONVENTIONAL — conventional metalic partial denture
  Other Names: partial denture
  Arms: conventional group

SUMMARY:
Purpose: Evaluation of patients' satisfaction, biting force measurement and radiographic evaluation of abutment teeth of tooth implant supported bridge, unilateral attachment and conventional partial denture in mandibular distal extension cases.

Materials and methods: Twenty four patients were selected and divided into three equal groups, each of eight patients: patients of group I Patients received a fixed tooth implant supported bridge, patients of group II Patients received a removable unilateral attachment partial denture and group III Patients received a conventional removable partial denture.Evaluation included patient satisfaction and biting force measurement radiographic evaluation of terminal abutments.

DETAILED DESCRIPTION:
Purpose: Evaluation of patients' satisfaction, biting force measurement and radiographic evaluation of abutment teeth of tooth implant supported bridge, unilateral attachment and conventional partial denture in mandibular distal extension cases.

Materials and methods: Twenty four patients were selected according to the following criteria: Patients with unilateral mandibular distal extension with last standing second premolar abutment, abutments showed sufficient occluso-gingival height and good periodontal condition. Patients were divided into three equal groups, each of eight patients: patients of group I Patients received a fixed tooth implant supported bridge, patients of group II Patients received a removable unilateral attachment partial denture and group III Patients received a conventional removable partial denture.Evaluation included patient satisfaction using "OHIP14" questionnaires and biting force measurement radiographic evaluation of terminal abutments.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral mandibular distal extension area
* The abutments showed sufficient occluso-gingival height of its clinical crown
* Adequate inter-arch space and no tempro-mandibular joint disorders.
* No para-functional habits,
* Full opposing arch or restored with acceptable fixed restoration
* Minimal bone height11 mm at the lower second molar area.

Exclusion Criteria:

*Insufficent bone height in posterior area of mandible

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-09-20 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
patient satisfaction | 1 month
  questionnaires

SECONDARY OUTCOMES:
biting force | 1 month
  measuring the biting force of the patients by sensor
radiographic evaluation | 1 month
  evaluation of alveolar bone loss

CONTACTS AND LOCATIONS:
Overall Officials: samira Ibrahim, prof, Principal Investigator — professor of prosthodontics
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No